CLINICAL TRIAL: NCT05815394
Title: 177Lu-labeled NY108 SPECT Imaging in Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS2023013
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-Anti-PSMA mAbs (Experimental)
  Interventions: Drug: 177Lu-labeled NY108

INTERVENTIONS:
Drug: 177Lu-labeled NY108 — Patients will receive a tracer (40-60ug) dose of 177Lu(28.5-31.5mCi) labelled NY108.

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 177Lu-labeled NY108 (177Lu-NY108) SPECT Imaging in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age 18-75, male;
3. Clinical diagnosis of prostate cancer with diagnostic criteria referencing biopsy and at least one metastasis;
4. Patients must be 68Ga-NY108 Positron Emission Tomography (PET)/Computed Tomography (CT) scan positive;
5. Patients must have received at least one NAAD (such as enzalutamide and/or abiraterone) and at least one paclitaxel regimen;
6. Progressive metastatic destructive resistant prostate cancer as determined by PCWG3 criteria;
7. An ECOG score of 0-2

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with severe systemic or localized infections or other serious coexisting diseases;
3. Patients with abnormal immune function or who have recently used immunosuppressive or booster agents including various vaccines, etc;
4. Patients with autoimmune diseases, including rheumatoid, etc;
5. Inadequately controlled arrhythmias, including atrial fibrillation:
6. Cardiac insufficiency (New York Heart Association (NYHA) work class criteria);
7. Uncontrolled hypertension;
8. Patients with a history of allergy or hypersensitivity to any component of the imaging agent, including antibodies;
9. Subjects positive for syphilis, HBV, HCV, FIIV;
10. Subjects of childbearing age who are unable to use effective contraceptive devices:
11. Patients with a history of mental illness or related medical conditions;
12. Patients who are unable or unavailable for SPECT/CT scanning;
13. Other subjects who, in the opinion of the investigator, are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 177Lu-Anti-PSMA mAbs(NY108) | 1 year
  Biodistribution of 177Lu-Anti-PSMA mAbs(NY108) evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 177Lu-SPECT scans will be reported.
Incidence of Treatment-Emergent Adverse Events | 1 year
  Safety will be assessed by evaluation of incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjing Yu, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No